CLINICAL TRIAL: NCT01080989
Title: The Sero-prevalence and Genetic Study for the Infectious Diseases and Metabolic Syndrome in Solomon Islands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KMUH-IRB-980096
Record Dates: First submitted 2009-08-30; First posted 2010-03-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2011-04

CONDITIONS: Flavivirus Infection; Alphavirus Infections; Malaria; Parasitic Disease; Leptospirosis; Hypertension; Metabolic Syndromes
Keywords: solomon islands; malaria; flavivirus; alphavirus; parasite; leptospirosis
MeSH Terms: conditions — Flavivirus Infections; Alphavirus Infections; Malaria; Parasitic Diseases; Leptospirosis; Hypertension; Metabolic Syndrome | interventions — Therapeutics; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- health screening and clinical diagnosis and treatment for p (Other): The study project can be divided into two parts: (1) health screening for the community and (2) clinical diagnosis and treatment for patients at National Referral Hospital (NRH) in Solomon islands.
  Interventions: Other: diagnosis, treatment and education

INTERVENTIONS:
Other: diagnosis, treatment and education — Drug:
  anti-intestinal parasitic drugs:
  1. mebendazole 500mg one dose (For Hook worm infections, Ascariasis, Trichuriasis)
  2. albendazole(400 mg bid * 7days) or Ivermectin(200 mcg/kg/day * 2 days) (For Strongyloidiasis).
  Behavior:
  1. Education capacity building (for local health personals): promote their ability of diagnosis and education to the community and patients for the associated diseases in this study.
  2. Assist the trained local health personals to educate the patients and the community from the design of teaching materials and the contents.

SUMMARY:
The study project can be divided into two parts: (1) health screening for the community and (2) clinical diagnosis and treatment for patients at National Referral Hospital (NRH) in Solomon islands. The health screening includes a questionnaire, stool parasitic screening and blood laboratory tests. A total of 800 subjects will participate in this study. The collected samples are venous blood (20 ml/per subject) and stool in order to conduct the related tests mentioned above.

As for the collection of target patients, KMUH will cooperate with NRH to collect two kinds of blood samples: the blood samples of confirmed malarial cases and those of cases suspicious of Flaviviral, Alpha-viral, Rickettsial, and Leptospiral infections. The expected received cases are 600 each year. The venous blood samples (20 ml/per subject) will be used to conduct related tests mentioned above. At the same time, the subjects will also have to fill out a related questionnaire which includes height, weight, waist line, heath behavior and habit, and past history, etc.

DETAILED DESCRIPTION:
KMUH plan a series of medical services to Solomon Islands with the expectation that the health and medical standard in Solomon Islands can be improved by medical interaction and the use of high-tech medical instruments. By collecting data from Solomon Islands, KMUH can better understand the health needs, the characteristics of diseases, and the basic health information of Solomon Islanders so that the strategies and the operation goals for further improvement will be more explicit for KMUH's medical teams.

The medical service and study project can be divided into two parts: (1) health screening for the community and (2) clinical diagnosis and treatment for patients at NRH. The health screening includes a questionnaire, stool parasitic screening and blood laboratory tests. In the questionnaire, height, weight, waist line, health behavior and habit, and past history are investigated. In the laboratory tests, parasite screening, Malaria rapid check, Flavivirus including dengue virus and Japanese virus, the seroprevalence of Rickettsia, HIV test, Diabetes, gout, cardiovascular risk factors, and fungal infection are included. A total of 800 subjects will participate in this study. The collected samples are venous blood (20ml/per subject) and stool in order to conduct the related tests mentioned above.

As for the collection of target patients, KMUH will cooperate with NRH in the Solomon islands to collect two kinds of blood samples: the blood samples of confirmed malarial cases and those of cases suspicious of Flaviviral, Rickettsial,and Leptospiral infections. The expected received cases are 600 each year. The blood samples of confirmed malarial cases will be used for pathogen identification and drug resistance analysis. The blood samples suspicious of Flaviviral(dengue virus, Japanese encephalitis virus), Alpha-viral(Chikungunya virus, Ross river virus), Rickettsial, and Leptospiral infections will be used for the following tests of either one, including ICT (immuno- chromatographic test) rapid test, ELISA, PCR (polymerase chain reaction) and the isolation and identification of pathogens. The venous blood samples (20ml/per subject) will be used to conduct related tests mentioned above. At the same time, the subjects will also have to fill out a related questionnaire which includes height, weight, waist line, heath behavior and habit, and past history, etc. For the confirmed malarial cases, the frequency of blood drawing will start from the diagnosed day, and the 3rd, the 7th , the 14th, the 21st , and the28th days after treatment, with total six times sampling. The blood samples will be used to identify malaria pathogen types and conduct drug resistance analysis.

ELIGIBILITY:
Inclusion Criteria:

1. For community participants: Health volunteers who are willing to join this study (including the stool and blood testing) after explanation and sign the informed consents.
2. For hospital cases: The patients ,who were suspicious of malaria, leptospirosis, Alpha-viral(Chikungunya virus, Ross river virus), and flavivirus infections (dengue fever, Japanese encephalitis..ect) by the attending physicians, will be informed about this study by drawing blood samples if they agree to participate.

Exclusion Criteria:

1. The participants whose stool or blood samples were in-adequate or missing will be excluded from this study.
2. The participants whose documented personal information is fake or cannot be identifiable will also be excluded from this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1477 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
health screening for the community | one per year
  Survey the prevalence of intestinal parasitic diseases, flaviviral(Dengue and Japanese encephalitis), Alpha-viral(Chikungunya virus, Ross river virus), leptospiral and malarial infections, and metabolic syndromes(hypertension, diabetes mellitus, hyperlipidemia and gout).

SECONDARY OUTCOMES:
Patients of confirmed malarial cases and those of cases suspicious of Flaviviral, Alpha-viral, Rickettsial,and Leptospiral infections. | one per year
  1. The confirmed malarial cases will be used for pathogen identification and drug resistance analysis. The cases suspicious of Flaviviral (dengue virus, Japanese encephalitis virus), Alpha-viral(Chikungunya virus, Ross river virus), Rickettsial, and Leptospiral infections will be used for the following tests of either one, including ICT (immuno- chromatographic test) rapid test, ELISA, PCR, and the isolation and identification of pathogens.
  2. Evaluate the incidence of above diseases after interventions(treatment, management and education capacity buildings).

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hsiung Sheu, Dr, Study Chair — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshiung, Taiwan